CLINICAL TRIAL: NCT04724304
Title: Myocardial Blood Volume Measurement by Real-Time Myocardial Perfusion Echocardiography Correlates to Myocardial Compressibility by Cardiac Magnetic Resonance Imaging in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Courtney E. Bennett, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20-000936
Record Dates: First submitted 2021-01-22; First posted 2021-01-26 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy adults (Experimental): Healthy adults will have blood flow to the heart evaluated using s Real-Time Myocardial Echocardiography (RTMPE) and magnetic resonance image (MRI) to the heart.
  Interventions: Diagnostic Test: Real-Time Myocardial Echocardiography (RTMPE); Diagnostic Test: Magnetic resonance image (MRI)

INTERVENTIONS:
Diagnostic Test: Real-Time Myocardial Echocardiography (RTMPE) — Uses sound waves (ultrasound) to produce an images of the heart. During RTMPE a microbubble contrast agent is administered through an intravenous line (IV) to make the images of your heart clearer.
Diagnostic Test: Magnetic resonance image (MRI) — Imaging that focuses on the heart or blood vessels to assess size and function of the heart's chambers, thickness and movement of the walls of the heart, and blood flow in the blood vessels.

SUMMARY:
This study is being done to find out the normal amount of blood within the heart muscle and the variations in this blood flow between a cardiac MRI and TTE.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Available for testing performed in Rochester, MN.
* Willing to undergo both an echocardiogram with RTMPE and CMR.
* Study subject providing consent.

Exclusion Criteria:

* Adults < 18 years.
* BMI <30 kg/m^2.
* Hypertension.
* Diabetes Mellitus.
* Stroke.
* Cardiomyopathy or structural heart disease.
* Known coronary artery disease or history of myocardial infarction.
* Contraindication to echo enhancement agent or gadolinium administration such as an allergy.
* Renal GFR < 50 mL/mL.
* Females who are pregnant.
* Subject unwilling to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Myocardial blood volume | Baseline
  Ratio in systole and diastole (MBVs/MBVd) by real-time myocardial perfusion echocardiography (RTMPE)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Bennett, D.O., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials